CLINICAL TRIAL: NCT03801759
Title: A Phase 1 Open-label, Three Arm Study in Healthy Adult Volunteers to Assess Vadadustat as a Perpetrator in Drug-Drug-Interactions With Digoxin, Adefovir and Furosemide
Brief Title: Drug-Drug Interaction Study of Vadadustat With Digoxin, Adefovir and Furosemide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: AKB-6548-CI-0031
Record Dates: First submitted 2018-12-27; First posted 2019-01-11 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Drug Interaction Potentiation
Keywords: vadadustat; drug interactions; healthy volunteers
MeSH Terms: interventions — vadadustat; Furosemide; adefovir; Digoxin

STUDY DESIGN:
Intervention Model Description: Each arm has fixed sequence design.
  1. Arm 1 (n = 20): Digoxin 0.5 mg alone, vadadustat 600 mg alone and digoxin + vadadustat
  2. Arm 2 (n = 16): adefovir 10mg alone, vadadustat 600 mg QD alone and adefovir + vadadustat
  3. Arm 3 (n=22) : furosemide 40mg alone, vadadustat 600 mg QD alone, and furosemide + vadadustat
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vadadustat, digoxin (Experimental): Arm 1: Subjects will receive a single oral dose of digoxin 0.5 mg alone, followed by a washout period and repeat doses of vadadustat 600 mg QD alone and in combination with a single dose of digoxin 0.5 mg.
  Interventions: Drug: Vadadustat; Drug: Digoxin
- Vadadustat, adefovir (Experimental): Arm 2: Subjects will receive a single dose of oral adefovir 10 mg alone, followed by a washout period and repeat doses of vadadustat 600 mg QD alone and in combination with a single dose of adefovir.
  Interventions: Drug: Vadadustat; Drug: Adefovir
- Vadadustat, Furosemide (Experimental): Arm 3: Subjects will receive a single dose of oral furosemide 40 mg alone, followed by a washout period and repeat doses of vadadustat 600 mg QD alone, and in combination with a single dose of furosemide 40 mg.
  Interventions: Drug: Vadadustat; Drug: Furosemide

INTERVENTIONS:
Drug: Vadadustat — Oral dose 600 mg
  Other Names: AKB 6548
Drug: Furosemide — Oral Furosemide
  Arms: Vadadustat, Furosemide
Drug: Adefovir — Oral Adefovir
  Arms: Vadadustat, adefovir
Drug: Digoxin — Oral Digoxin
  Arms: Vadadustat, digoxin

SUMMARY:
This is a Phase 1, open-label, 3-arm, fixed sequence, study to evaluate vadadustat as a perpetrator of drug-drug interactions (DDIs) with digoxin, adefovir and furosemide in healthy male and female subjects.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, 3-arm, fixed sequence, study to evaluate vadadustat as a perpetrator of drug-drug interactions (DDIs) with digoxin, adefovir and furosemide in healthy male and female subjects. Unique subjects will be enrolled into each arm of the study and enrollment will be sequential. The first 20 subjects confirmed to be eligible will be assigned to Arm 1 (digoxin), the next 16 subjects will be assigned to Arm 2 (adefovir) and the next 22 subjects will be assigned to Arm 3 (furosemide). Blood samples for PK analysis will be collected at pre-defined timepoints for each arm throughout the study. Subjects will be on study for up to 80 days, including a 28-day screening period, 7-21 day in clinic period, and a 30-day follow up period post last dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male or female between 18 and 55 years of age, inclusive, at time of informed consent.
* Body mass index between 18.0 and 30.0 kg/m2, with a minimum body weight of 45 kg for females and 50 kg for males, inclusive.

Exclusion Criteria:

* Current or past clinically significant history of cardiovascular, cerebrovascular, pulmonary, gastrointestinal, hematologic, renal, hepatic, immunologic, metabolic, urologic, neurologic, dermatologic, psychiatric, or other major disease. History of cancer (except treated non-melanoma skin cancer) or history of chemotherapy use within 5 years prior to Screening.
* Positive test results for human immunodeficiency virus (HIV) antibody; Positive test results of hepatitis B surface antigen (HBsAg), or positive hepatitis C virus antibody (HCVab) within 3 months prior to screening; or positive test results for human immunodeficiency virus antibody (HIVab) at Screening
* Taking any prescription medication or over the counter multi-vitamin supplement, or any non-prescription products (including herbal-containing preparations but excluding acetaminophen) within 14 days prior to Day -1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from 0 to last quantifiable concentration (AUClast) for digoxin, adefovir and furosemide | Up to 12 Weeks
Area under plasma concentration-time curve from 0 to infinity (AUCinf) for digoxin, adefovir and furosemide | Up to 12 Weeks
Maximum observed plasma concentration (Cmax) for digoxin, adefovir and furosemide | Up to 12 Weeks

SECONDARY OUTCOMES:
Time to maximum observed plasma concentration (Tmax) for digoxin, adefovir and furosemide | Up to 12 Weeks
Elimination rate constant (Kel) for digoxin, adefovir and furosemide | Up to 12 Weeks
Terminal half-life (t½) for digoxin, adefovir and furosemide | Up to 12 Weeks
Apparent total body clearance (CL/F) for digoxin, adefovir and furosemide | Up to 12 Weeks
Percent of extrapolated area under the curve from time t to infinity (%AUCextrap) for digoxin, adefovir and furosemide | Up to 12 Weeks
Reporting of Treatment Emergent Adverse Events (TEAEs) as reported by study subjects | Up to 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Akebia Therapeutics, Study Director — Sponsor GmbH
Locations (1):
- inVentiv Health Clinique Inc., Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided